CLINICAL TRIAL: NCT03938142
Title: Goalsetting in Patients With Chronic Pain: a European Survey
Status: Completed | Type: Observational
Sponsor: Moens Maarten (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: Goalsetting
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with chronic pain
  Interventions: Other: Filling in an online survey regarding goalsettings

INTERVENTIONS:
Other: Filling in an online survey regarding goalsettings — Patients are asked to fill in an online survey regarding their individual goalsettings.

SUMMARY:
The aim of this survey is to get insight in the individual goals of chronic pain patients according to the ICF framework.

ELIGIBILITY:
Inclusion Criteria:

* patients who are suffering from chronic pain

Exclusion Criteria:

* healthy participants or patients with acute pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 1494 (Actual)
Dates: Start 2019-11-23 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Individual goalsettings | at the moment of filling in the survey (cross-sectional)
  Individual goals that patients want to achieve with their treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium